CLINICAL TRIAL: NCT00114634
Title: Short-Term Behavioral Effects of Cholesterol Therapy in Smith-Lemli-Opitz Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Forbes Porter, M.D., Senior Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 050168; 05-CH-0168 (Other: NIH CC)
Record Dates: First submitted 2005-06-15; First posted 2005-06-16 (Estimated); Results first posted 2014-04-09 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2015-12

CONDITIONS: Smith-Lemli-Opitz Syndrome
Keywords: SLOS; RSH syndrome; ABC Checklist; Cholesterol supplementation; Egg yolk; Smith-Lemli-Opitz Syndrome
MeSH Terms: conditions — Smith-Lemli-Opitz Syndrome | interventions — Cholesterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Egg yolk preparation with cholesterol (Experimental): Dietary cholesterol in the form of liquid egg yolk
  Interventions: Dietary Supplement: Egg yolk preparation with cholesterol
- Egg yolk preparation without cholesterol (Placebo Comparator): No dietary cholesterol supplementation (egg substitute) Papetti Foods "Better 'n Eggs" egg substitute
  Interventions: Dietary Supplement: Egg substitute, without cholesterol

INTERVENTIONS:
Dietary Supplement: Egg yolk preparation with cholesterol — Egg yolk preparation with cholesterol
  Arms: Egg yolk preparation with cholesterol
Dietary Supplement: Egg substitute, without cholesterol — Placebo control. Egg substitute, without cholesterol
  Arms: Egg yolk preparation without cholesterol

SUMMARY:
This 10-week study will evaluate and compare behavior changes in children with Smith-Lemli-Opitz syndrome (SLOS) who are taking cholesterol supplementation versus those who are not on cholesterol supplementation. SLOS is a genetic disorder that affects the development of children both before and after birth. An enzyme deficiency in these children results in low levels of cholesterol, which can cause a variety of birth defects and behavioral problems. Typical abnormal physical features of patients include a small head, drooping eyelids, small upturned nose, small chin, cleft palate, heart defects, and extra fingers or toes.

Children between 5 and 17 with mild SLOS who do not have a history of egg allergy or intolerance may be eligible for this study. Candidates are screened with a questionnaire about the patient's age, genotype (if known), sterol levels, symptoms, current treatment and medical history.

Children participate in two 2-week study phases. Between the study phases the children will take 150 mg/kg daily of a cholesterol preparation typically used to supplement cholesterol in patients in SLOS studies at NIH. In the study phases, the participants are randomly assigned to take either egg yolk or an egg yolk substitute, such as Egg Beaters, that does not contain cholesterol. The study is done at the participant's home, and the cholesterol supplementation and egg/egg substitute are sent to the home each day with instructions on how to take them.

The caretakers can stop the study phases after four days if behavior problems occur.

The children's caretakers fill out a standard behavioral questionnaire, the Aberrant Behavior Checklist. The questionnaire is designed to assess the effects of treatment in mentally impaired persons.

DETAILED DESCRIPTION:
Smith-Lemli- Opitz syndrome (SLOS) is an autosomal recessive genetic condition caused by a deficiency of the enzyme 3beta-hydroxysterol delta(7)- reductase (DHCR7). DHCR7 is the final enzyme in the sterol synthetic pathway and converts 7- dehydrocholesterol (7DHC) to cholesterol. This results in low cholesterol and elevated 7DHC levels. SLOS has a wide phenotypic spectrum. Mildly affected individuals may have subtle dysmorphic features along with learning and behavioral disabilities. Typical clinical manifestations include microcephaly, ptosis, anteversion of the nostrils, micrognathia, high arched or cleft palate, congenital heart defects, clinodactyly, post- axial polydactyly, and 2-3 toe syndactyly. More severely affected individuals have multiple congenital anomalies, may be miscarried, stillborn, or die within the first few weeks of life.

Dietary cholesterol supplementation in children with SLOS is reported to improve behavior, growth and nutritional status. Based upon observational studies, the behavioral changes reported with dietary cholesterol supplementation occur rapidly and appear to be reversible. Parental reports of improved behavior could be influenced by a placebo effect. Thus, we are proposing a blinded study to compare behavioral changes while the patient is on cholesterol supplementation (egg yolk) versus no cholesterol supplementation (egg substitute).

The objectives of this study are:

1. To quantitatively evaluate behavior, in a blinded study, of SLOS children on and off dietary cholesterol supplementation.
2. To quantitatively evaluate behavior in SLOS children treated with egg yolk compared to synthetic dietary cholesterol supplementation.

Completed study has been published. Tierney, E., Conley, S.K., Goodwin, H., Porter, F.D. (2010) Analysis of short-term behavioral effects of dietary cholesterol supplementation in Smith-Lemli-Opitz Syndrome. Am. J. Med. Genet. Part A. 152A: 91-95 PMID: 20014133

ELIGIBILITY:
Inclusion

1. This study will include pediatric patients, ages 4-17 years old with a biochemical diagnosis of Smith-Lemli-Opitz Syndrome (SLOS).
2. Only mild and classical patients will be enrolled.
3. This study will be open to include SLOS patients regardless of whether or not they are participating in another NIH protocol.

Exclusion

1. Patients with a history of egg allergy or intolerance will be excluded from this study.
2. Subjects must be well enough to be in a home setting.
3. Patients participating in our simvastatin protocol (03-CH-3225) will be excluded from this study.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2005-06; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Forbes D Porter, MD, Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Elias ER, Irons MB, Hurley AD, Tint GS, Salen G. Clinical effects of cholesterol supplementation in six patients with the Smith-Lemli-Opitz syndrome (SLOS). Am J Med Genet. 1997 Jan 31;68(3):305-10. doi: 10.1002/(sici)1096-8628(19970131)68:33.0.co;2-x. PMID 9024564
- [Background] Irons M, Elias ER, Abuelo D, Bull MJ, Greene CL, Johnson VP, Keppen L, Schanen C, Tint GS, Salen G. Treatment of Smith-Lemli-Opitz syndrome: results of a multicenter trial. Am J Med Genet. 1997 Jan 31;68(3):311-4. PMID 9024565
- [Background] Kelley RI. A new face for an old syndrome. Am J Med Genet. 1997 Jan 31;68(3):251-6. doi: 10.1002/(sici)1096-8628(19970131)68:33.0.co;2-p. No abstract available. PMID 9024554

RESULTS

PARTICIPANT FLOW:
Recruitment Details: October to July 2008
Pre-assignment Details: no exclusions
Groups:
- Egg Yolk or no Egg Yolk: This was a double-blind, placebo-controlled, cross-over design. The trial was composed of five 2-week phases. Two phases, phases 2 and 4, were double-blinded. During these phases, subjects were either on placebo (egg substitute with no cholesterol) or cholesterol supplementation (pasteurized egg yolk). During the interval phases, 1, 3 and 5, subjects were maintained on baseline therapy of 150 mg/kg/day of crystalline cholesterol suspended in Ora-Plus. Order of placebo versus cholesterol was random with 6 subjects receiving placebo first (in phase 2) and 4 subjects receiving cholesterol containing pasteurized egg yolk first. 13 subjects were enrolled, only 10 subjects completed the study.
Period: Overall Study
Arm/Group | Egg Yolk or no Egg Yolk
Started | 13
Completed | 10 (Assessment forms lost by one failure to complete and return forms by two)
Not Completed | 3
Not completed — failure to return forms | 3

BASELINE CHARACTERISTICS:
Groups:
- Egg Yolk or no Egg Yolk: All subjects were on cholesterol suspension or egg yolk versus no egg yolk.
Arm/Group | Egg Yolk or no Egg Yolk
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.4 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 10
Severity score [Median (Full Range); unit: units on a scale] — Severity score ranges from 0-100; the higher the score the greater the severity
  units on a scale | 17 [6 to 28]

OUTCOME MEASURES:

1. Primary Outcome: Hyperactivity Sub-scale of the Aberrant Behavior Checklist-Community (ABC-C).
Description: The Aberrant Behavior Checklist-Community (ABC-C) is a measure used to identify treatment efficacy among intellectually impaired individuals. ABC Subscale IV (Hyperactivity) has 16 items, each can be rated from 0 to 3, with 0 equal to not at all a problems, one the problem is the behavior but slight in degree, to the problem is moderately serious, 3 the problem is severe in degree. For this subscale, score can go from 0 - 48. The higher the score, the worse the hyperactivity. The comparison in this study was made between the blinded phases when patients received either egg yolk (treated, +cholesterol) or egg substitute (untreated, -cholesterol). Order was randomized.
Time Frame: 2 weeks
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Crossover Study: This was a double-blind, placebo-controlled, cross-over design. The trial was composed of five 2-week phases. Two phases, phases 2 and 4, were double-blinded. During these phases, subjects were either on placebo (egg substitute with no cholesterol) or cholesterol supplementation (pasteurized egg yolk). During the interval phases, 1, 3 and 5, subjects were maintained on baseline therapy of 150 mg/kg/day of crystalline cholesterol suspended in Ora-Plus. Order of placebo versus cholesterol was random with 6 subjects receiving placebo first (in phase 2) and 4 subjects receiving cholesterol containing pasteurized egg yolk first. 13 subjects were enrolled, only 10 subjects completed the study.
Arm/Group | Crossover Study
Number analyzed (Participants) | 10
units on a scale
  Untreated | 8.6 (2.3)
  Treated | 8.6 (2.2)
Statistical Analysis 1: Comparison: Crossover Study; Test type: Superiority or Other; p = 1.0, t-test, 2 sided

2. Secondary Outcome: ABC Irritability Sub-scale
Description: ABC Subscale I (Irritability) has 15 items, each can be rated from 0 to 3, with 0 equal to not at all a problem, 1 the problem is the behavior but slight in degree, 2 the problem is moderately serious, 3 the problem is severe in degree. For this subscale, score can go from 0 - 45
Time Frame: 2 weeks
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Placebo: egg substitute
- Cholesterol: pasteurized egg yolk
Arm/Group | Placebo | Cholesterol
Number analyzed (Participants) | 10 | 10
units on a scale | 8.300 (2.2) | 8.8 (1.9)

3. Secondary Outcome: ABC Lethargy Sub-scale
Description: ABC Subscale II (Lethargy) has 16 items, each can be rated from 0 to 3, with 0 equal to not at all a problems, 1 the problem is the behavior but slight in degree,2 the problem is moderately serious, 3 the problem is severe in degree. For this subscale, score can go from 0 - 48.
Time Frame: 2 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Cholesterol
Number analyzed (Participants) | 10 | 10
units on a scale | 3.7 (0.7) | 3.6 (0.8)

4. Secondary Outcome: ABC Stereotypy Sub-scale
Description: ABC Subscale III (Stereotypy) has 7 items, each can be rated from 0 to 3, with 0 equal to not at all a problems, 1 the problem is the behavior but slight in degree, 2 the problem is moderately serious, 3 the problem is severe in degree. For this subscale, score can go from 0 - 21.
Time Frame: 2 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Cholesterol
Number analyzed (Participants) | 10 | 10
units on a scale | 1.6 (0.6) | 2.0 (0.8)

5. Secondary Outcome: ABC Inappropriate Behavior Sub-scale
Description: ABC Subscale V (Inappropriate speech) has 4 items, each can be rated from 0 to 3, with 0 equal to not at all a problems, 1 the problem is the behavior but slight in degree, 2 the problem is moderately serious, 3 the problem is severe in degree. For this subscale, score can go from 0 - 12.
Time Frame: 2 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Cholesterol
Number analyzed (Participants) | 10 | 10
units on a scale | 1.0 (0.4) | 1.0 (0.4)

6. Secondary Outcome: ABC Total Score
Description: ABC total score includes all the questions from subscales, with range of 0 to 174. Higher the score , the greater the problem.
Time Frame: 2 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Cholesterol
Number analyzed (Participants) | 10 | 10
units on a scale | 23.2 (4.8) | 23.0 (3.2)

ADVERSE EVENTS:
Groups:
- Group 1: All subjects were on cholesterol suspension or egg yolk versus no egg yolk.
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

LIMITATIONS AND CAVEATS:
Poor power due to low enrollment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No